CLINICAL TRIAL: NCT00884000
Title: A Randomised, Open-label, Parallel-group, Multi-centre Trial to Compare the Efficacy and Safety for 12 Months of Zomacton to Genotropin in Children With Idiopathic Growth Hormone Deficiency
Brief Title: A Study of Zomacton in Children With Growth Hormone Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE999905 CS07; 2008-004849-28
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Genotropin
- 2 (Experimental)
  Interventions: Drug: Zomacton

INTERVENTIONS:
Drug: Genotropin
  Arms: 1
Drug: Zomacton
  Arms: 2

SUMMARY:
This trial is set up to compare Zomacton to Genotropin for the treatment of growth hormone deficiency in children. The children will be treated for 1 year. Half of the patients will be treated with Genotropin and half with Zomacton. During this time they will be dosed every day by themselves or their parents at home in the evening. There will be 138 patients in the trial from age 3 to age 11. The patients cannot have been treated before with growth hormone and the patients must have a proven growth hormone deficiency, this will be shown by a specific test that will be performed before the trial in the local clinic and once during the trial. During the time of the treatment the patients will come to visit the clinic every 3 months. At these visits their heights will be measured, blood samples will be taken, physical examinations will be performed and questions about their health will be asked. At 2 times in the trial they will have a hand x-ray taken to measure the bone age. At the end of the trial the patients will stop the treatment and continue on one of the marketed products available to treat growth hormone deficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Children aged ≤3yrs old and not above 10 yrs for girls or 11 yrs for boys
3. Idiopathic growth hormone deficiency confirmed during the pre-screening period by a standard GH stimulation test (defined as peak level of <10ng/ml pr lower if so required by the country specific board(s)
4. Height SDS <-2 SD of ref value for CA
5. Height velocity SDSCA ≤ 0 SD of ref value for at lease 6 months prior to pre-screening
6. Height recorded for at least 6 months but not more than 18 months of pre-screening
7. The difference between CA-BA≥ 1
8. A positive locally performed GH stimulation test (defined as a peak plasma level of<9ng/ml or lower if so required by the country specific board(s)) prior to the pre-screening

Exclusion Criteria:

1. BA above 9 yrs for girls and 10 yrs for boys
2. Puberty Tanner stage >1
3. Weight <12 Kg at screening
4. Any prior treatment with GH
5. Closed epiphysis
6. Any diagnosed or suspected syndrome (e.g. Silver -Russell, Turner's or seckel syndrome) which possibly could affect growth
7. Any other diagnosed or suspected endocrine or metabolic disorder
8. Any diagnosed or suspected sever chronic disease
9. Clinical signs of dysmorphic features, malformations or mental retardations
10. Growth failure due to other disorders
11. Previous or present use of drugs that could interfere with GH treatment (e.g. steroids)
12. Diagnosed malignant disease
13. Any abnormal CS lab results that requires further investigation
14. Receipt of an investigational drug within the last 28 days preceding screening or longer if considered possible to influence the outcome of the current trial
15. Any knowledge of hypersensitivity to somatropin or any of the excipients of Zomacton or Genotropin

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 165 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Height Velocity | 12 months

SECONDARY OUTCOMES:
Height SDS | 12 months
Height velocity SDS | 12 months
Change in IGF-1 and IGFBP-3 | 12 months
BA (Bone Age) | 12 months
Anti-hGH AB | 12 months
AE and tolerability | 12 months
CS Changes in safety lab, physical examination and vital signs | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (43):
- Hungary (5):
  - Semmelweiss University, 1st dept of paediatrics, Budapest
  - Szent Janos Kh Budai, Budapest
  - Petz Country Teaching Hospital, Győr
  - University of Szeged, Szeged
  - Markusovszkty Teaching Hospital, Szombathely
- India (8):
  - Associates in Clinical Endocrinology Education and Research (ACEER), Chennai
  - Apollo Hospitals, Hyderabad
  - TOTALL Diabetes Hormone Institute, Indore
  - KEM Hospital, Mumbai
  - Prince Aly Khan Hospital, Mumbai
  - Endocare Clinic, Nashik
  - Jehangir Clinical Development Centre Pvt. Ltd., Jehangir Hospital, Pune
  - Health & Research Centre, Trivandrum
- Israel (7):
  - Haemek Medical Center, Afula
  - Soroka University Medical Center, Beersheba
  - Western Galilee Medical Center, Nahariya
  - Schneider Children's Medical Center of Israel, Petah Tikva
  - Edmond and Lily Safra Children's hospital - The Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Dana Children's Hospital - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Poland (4):
  - Wojewódzki Szpital Dziecięcy im. J.Brudzińskiego w Bydgoszczy, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdańsk, Gdansk
  - Uniwersytecki Szpital Dziecięcy w Krakowie, Krakow
  - SPSK nr.1 im. Prof. T. Sokołowskiego PAM Szczecin, Szczecin
- Romania (6):
  - Societatea Civila Medicala "Dr. Paveliu", Bucharest
  - Spitalul Clinic Municipal "Filantropia", Craiova
  - Spitalul Clinic Judetean de Urgenta "Sf. Spiridon", Iași
  - Spitalul Clinic Judetean Mures, Târgu Mureş
  - Paediatric Endocrinology/Medicali's SRL, Timișoara
  - Spitalul Clinic pentru Copii Louis Turcanu, Timișoara
- Russia (6):
  - State Educational Institution of Higher Professional Education "Kazan State Medical University of ROSZDRAV, Kazan'
  - Federal State Institution, Moscow
  - Russian Medical Academy of Post-graduate Education, Moscow
  - Saint-Petersburg State Health Care Institution, Saint Petersburg
  - State Educational Institution for Higher Professional Education, Saratov
  - State Educational Institution of Higher Professional Education "Siberian State Medical University of ROSZDRAV, Tomsk
- Ukraine (7):
  - Donetsk Regional Clinical Children's Hospital, Donetsk
  - Ivano-Frankivsk Regional Children Clinical Hospital, Ivano-Frankivsk
  - Kharkiv Regional Clinical Children's Hospital, Kharkiv
  - Institute of Endocrinology and Metabolism, Kiev
  - Ukrainian Children's Specialized Clinical Hospital, Kiev
  - Odessa National Medical University - (Located at Odessa Region Children's Clinical Hospital), Odesa
  - Zaporizhzhya Regional Paediatric Hospital, Zaporizhya